CLINICAL TRIAL: NCT03127072
Title: A Prospective, Randomized, One-center Study Assessing Overall Survival Using RFA Plus Chemotherapy ± Target Therapy and Chemotherapy ± Target Therapy Alone in Patients With Unresectable Unresectable Colorectal Cancer Liver Metastases
Brief Title: Study Comparing Radio Frequency Ablation Plus Chemotherapy and Chemotherapy Alone in Patients With Unresectable CRLM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Prof., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFACRLM
Record Dates: First submitted 2017-04-19; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer Liver Metastasis
Keywords: colorectal cancer; liver metastasis; Radiofrequency Ablation; chemotherapy; target therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): RFA plus chemotherapy ± target therapy
  Interventions: Device: Radiofrequency Ablation (RFA); Drug: chemotherapy ± target therapy
- Arm B (Active Comparator): chemotherapy ± target therapy
  Interventions: Drug: chemotherapy ± target therapy

INTERVENTIONS:
Device: Radiofrequency Ablation (RFA) — The radiofrequency generator has the capacity to deliver 200 watts of alternating current to the needle electrode for the coagulation necrosis of soft tissue
  Arms: Arm A
Drug: chemotherapy ± target therapy — chemotherapy ± target therapy

SUMMARY:
To date no prospective trials have been completed that demonstrated whether RFA is an effective adjunct to systemic chemotherapy (target therapy) with respect to advantages in overall survival compared with chemotherapy (target therapy) alone. The primary objective of this trial is to determine overall survival for patients with colorectal cancer liver metastasis are treated with radiofrequency ablation plus chemotherapy ± target therapy, compared to chemotherapy ± target therapy only.

ELIGIBILITY:
Inclusion Criteria:

All patients must meet the following criteria:

Patients must have incurable CRLM

Patients must have no more than 10 liver metastases (LMs) remaining after surgical resection, with diameter less than 5cm

Patients is medically eligible to receive RFA, as determined by the MDT (multidisciplinary team)

Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1

Age > 18 years

Subject life expectancy > 3 months

Platelets > 100×103/mm3

Total bilirubin <1.5mg/dl

Creatinine level < 2.0 mg/dl

All patients must sign an informed consent form

Exclusion Criteria:

The CRLM is amenable to curative surgical therapy

Uncorrectable coagulopathy

Subject is pregnant, nursing, or wishes to become pregnant during the study

Other serious medical condition (uncontrolled infection, uncontrolled cardiac disease) would preclude study treatment or impact survival

Current or planned treatment with any experimental chemotherapy or target drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-04-30 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival in subjects receiving RFA plus chemotherapy ± target therapy compared to chemotherapy ± target therapy alone was assessed from the date of study entry until death from the disease. | 3 years

SECONDARY OUTCOMES:
The differences in the incidence or severity of adverse events in the RFA plus chemotherapy ± target therapy arm compared to the chemotherapy ± target therapy only arm were was assessed by of complications after therapy. | 30 days post therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, PhD, Study Chair — Fudan University
Locations (1):
- Zhongshan hosptial, Fudan University, Shanghai, China